CLINICAL TRIAL: NCT07081360
Title: Neoadjuvant Chemotherapy Followed by Surgery Versus Upfront Surgery for Clearly Resectable Pancreatic Head Cancer and Periampullary Cancer: A Randomized Controlled Trial
Brief Title: Neoadjuvant vs Upfront Surgery for Resectable Pancreatic Cancer and Periampullary Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Saleh Khairy Saleh MD, Lecturer, Minia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1563/06/2025
Record Dates: First submitted 2025-07-04; First posted 2025-07-23 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Pancreas Cancer; Periampullary Cancer; Periampullary Carcinoma Resectable; Pancreatic Cancer Resectable; Ampullary Cancer; Pancreas Adenocarcinoma
Keywords: Pancreatic cancer; Neoadjuvant chemotherapy; Pancreaticoduodenectomy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Intervention Model Description: Two parallel groups: neoadjuvant chemotherapy followed by surgery versus upfront surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neoadjuvant chemotherapy group (mFOLFIRINOX) (Experimental): Neoadjuvant chemotherapy(mFOLFIRINOX) followed by pancreaticoduodenectomy
  Interventions: Drug: Neoadjuvant chemotherapy
- Upfront Surgery Group (Active Comparator): Pancreaticoduodenectomy followed by adjuvant chemotherapy
  Interventions: Procedure: Upfront Surgery Group

INTERVENTIONS:
Drug: Neoadjuvant chemotherapy — Neoadjuvant chemotherapy (mFOLFIRINOX) followed by pancreaticoduodenectomy
  Arms: Neoadjuvant chemotherapy group (mFOLFIRINOX)
Procedure: Upfront Surgery Group — Pancreaticoduodenectomy followed by adjuvant chemotherapy
  Arms: Upfront Surgery Group

SUMMARY:
Adjuvant chemotherapy after surgery significantly improved the survival of pancreatic cancer (PC) patients, but there is a problem that only about 50% of patients start adjuvant chemotherapy after pancreatectomy. Neoadjuvant chemotherapy might control potential metastatic lesions which are not being detected in early disease status and improve the R0 resection rate. In addition, it prevents futile surgery by selecting patients with rapid progression of disease. Furthermore, compared to chemotherapy administered after surgery, more patients can complete the planned chemotherapy schedule in neoadjuvant setting.

There are still few studies worldwide that prospectively explored the efficacy of neoadjuvant chemotherapy in resectable PC and periampullary cancer and the administration of neoadjuvant therapy in resectable PC depends on individual clinical judgment. Therefore, systematic and prospective clinical trials are essential to standardize treatment protocol in resectable PC and periampullary Cancer.

This randomized controlled trial compares neoadjuvant chemotherapy followed by surgery versus upfront surgery for patients with clearly resectable pancreatic head cancer and periampullary cancer. The study aims to determine if neoadjuvant chemotherapy improves overall survival compared to immediate surgery followed by adjuvant chemotherapy.

DETAILED DESCRIPTION:
Pancreatic cancer is the seventh highest cause of death from cancer worldwide, with only 20% of patients presenting with resectable disease. Despite potentially curative resections, 5-year survival remains at 20%. This study evaluates whether neoadjuvant chemotherapy can improve outcomes by eliminating occult metastatic disease and improving resection margins.

Patients with clearly resectable pancreatic head cancer or periampullary cancer will be randomized 1:1 to either neoadjuvant chemotherapy followed by open or laparoscopic pancreaticoduodenectomy (Arm A) or upfront laparoscopic pancreaticoduodenectomy followed by adjuvant chemotherapy (Arm B). The primary endpoint is overall survival, with secondary endpoints including R0 resection rate , disease-free survival and perioperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed pancreatic head cancer or periampullary carcinoma(endoscopic ultrasound (EUS)-guided biopsy).
* Clearly resectable disease as defined by National Comprehensive Cancer Network (NCCN) criteria on cross-sectional imaging:

No involvement or abutment of the celiac artery, common hepatic artery, superior mesenteric artery, or replaced right hepatic artery .

Less than 180 degree interface between tumor and vessel wall of the portal vein or superior mesenteric vein, and patent portal vein/splenic vein confluence No evidence of metastatic disease.

* Eastern Cooperative Oncology Group (ECOG)=0-1 & American Society of Anesthesiologists (ASA) score <4.
* Written informed consent.
* Medical history without previous pancreatic resection or pancreatic cancer.
* Adequate organ function (liver, kidney, bone marrow) (serum creatinine ≤2.0 mg/dL,reference range 0.5-1.20 mg/dL; serum albumin ≥2.5 g/dL, reference range 3.5-5.3; aspartate aminotransferase (AST) ≤95 U/L, reference range 0-38; Alanine aminotransferase (ALT) ≤102 U/L, reference range 0-41; prothrombin time ≤1.8, reference range 0-1.20; partial thromboplastin time ≤1.8, reference range 0.82-1.25; leukocyte count greater than 3.5×109/L, reference range 4.2-9.0; platelet count greater than 100×109/L, reference range 130-400; hemoglobin ≥9 g/dL, reference range 12-16).

Exclusion Criteria:

* Borderline resectable or locally advanced pancreatic or periampullary cancer.
* Tumor at the body or tail of the pancreas.
* Distant metastases.
* Prior chemotherapy , surgery or radiotherapy for pancreatic cancer.
* Severe comorbidities precluding surgery or chemotherapy.
* Pregnancy or lactation.
* Other neoplastic diseases (malignant)diagnosed in the past 5 years.
* Major surgery or traumatic event in the past 28 days.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Estimated)
Dates: Start 2025-07-20 (Actual); Primary Completion 2028-07-20 (Estimated); Study Completion 2028-08-20 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate | Up to 3 years.
  Overall survival will be measured as the time between date of randomization and date of death from any cause or date of last follow-up if alive.

SECONDARY OUTCOMES:
Disease-free survival (DFS) | Up to 3 years post-procedure.
  Disease-free survival will be measured as the time between date of surgery and date of disease recurrence
Local recurrence rate | Up to 3 years post-procedure.
  Local recurrence is defined as recurrence in the pancreatic resection margin, residual pancreas, and regional lymph nodes.The local recurrence is defined as the percentage of patients who had recurrence after the surgical resection.
Recurrence rate | Up to 3 years post-procedure.
  The proportion of patients who experienced recurrence within 3 years from the date of surgery.
Time to locoregional recurrence (TLR) | Up to 3 years post-procedure.
  Time to locoregional recurrence (TLR) is defined as the time from date of surgery to the date of locoregional recurrence after resection.
Response rate in neoadjuvant setting | 12 to 16 weeks.
  Defined as the percentage of patients who showed complete response, partial response, and stable disease after the scheduled neoadjuvant chemotherapy. The evaluation is based on RECIST v.1.1.
Time to distant metastases (TDM) | Time between randomization and metastases prior to surgery, metastases detected during surgery, or distant recurrence after resection, assessed up to 3 years.
  Time to distant metastases (TDM) is defined as the time from randomization to the date of metastases prior to surgery, metastases detected during surgery, or distant recurrence after resection.
Resection rate | At time of surgery or planned time of surgery.
  Referred to the proportion of patients who underwent curative resection
R0 resection rate | One to two weeks postsurgery.
  The percentage of patients that underwent a microscopically margin-negative (R0) resection. The resection is considered R0 if there is no tumor within 1 mm of the margins.
Lymph node-negative (N0) resection rate | One to two weeks postsurgery.
  The percentage of patients that underwent a resection with negative lymph nodes (N0) in the surgical specimen.
Pathologic complete response (pCR) rate | One to two weeks postsurgery.
  The rate (percentage) of patients who achieve a pathologic complete response (pCR) confirmed by histopathologic review of the surgical specimen.
Biomarker Response during neoadjuvant chemotherapy . | Baseline level is measured before start of neoadjuvant chemotherapy( within 1 week) , then after neoadjuvant therapy completion( 12 to 16 weeks).
  Carbohydrate antigen (CA) 19-9 levels predictive of response to neoadjuvant chemotherapy .
Rate of unresectability | At time of surgery or planned time of surgery.
  The rate (percentage) of patients who cannot undergo surgery due to adverse events, progressive disease, death, poor performance, or patient/physician decision, are deemed unresectable before surgery, or resection was not performed during surgery.
Chemotherapy start rate | upto 4 months.
  The percentage of patients who received at least one cycle of scheduled chemotherapy.
Number of chemotherapy cycles received. | up to 4 months.
  The number of scheduled chemotherapy cycles that patients received.
Chemotherapy completion rate | up to 4 months.
  The percentage of patients who completed all cycles of scheduled chemotherapy.
Perioperative Complications | From surgery until 90 days post-surgery
  The specific postoperative complications of pancreatic surgery include postoperative pancreatic fistula, postoperative hemorrhage ,bile leak and gastroparesis. Other common postoperative complications include abdominal infection, incision nonunion and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Saleh K Saleh, MD, Principal Investigator — Minia University
Locations (1):
- Liver and GIT hospital , Minia University, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Evans DB. The Complexity of Neoadjuvant Therapy for Operable Pancreatic Cancer: Lessons Learned From SWOG S1505. Ann Surg. 2020 Sep 1;272(3):487. doi: 10.1097/SLA.0000000000004131. No abstract available. PMID 32657915
- [Background] Murphy JE, Wo JY, Ryan DP, Jiang W, Yeap BY, Drapek LC, Blaszkowsky LS, Kwak EL, Allen JN, Clark JW, Faris JE, Zhu AX, Goyal L, Lillemoe KD, DeLaney TF, Fernandez-Del Castillo C, Ferrone CR, Hong TS. Total Neoadjuvant Therapy With FOLFIRINOX Followed by Individualized Chemoradiotherapy for Borderline Resectable Pancreatic Adenocarcinoma: A Phase 2 Clinical Trial. JAMA Oncol. 2018 Jul 1;4(7):963-969. doi: 10.1001/jamaoncol.2018.0329. PMID 29800971
- [Background] Golcher H, Brunner TB, Witzigmann H, Marti L, Bechstein WO, Bruns C, Jungnickel H, Schreiber S, Grabenbauer GG, Meyer T, Merkel S, Fietkau R, Hohenberger W. Neoadjuvant chemoradiation therapy with gemcitabine/cisplatin and surgery versus immediate surgery in resectable pancreatic cancer: results of the first prospective randomized phase II trial. Strahlenther Onkol. 2015 Jan;191(1):7-16. doi: 10.1007/s00066-014-0737-7. Epub 2014 Sep 25. PMID 25252602
- [Background] Casadei R, Di Marco M, Ricci C, Santini D, Serra C, Calculli L, D'Ambra M, Guido A, Morselli-Labate AM, Minni F. Neoadjuvant Chemoradiotherapy and Surgery Versus Surgery Alone in Resectable Pancreatic Cancer: A Single-Center Prospective, Randomized, Controlled Trial Which Failed to Achieve Accrual Targets. J Gastrointest Surg. 2015 Oct;19(10):1802-12. doi: 10.1007/s11605-015-2890-4. Epub 2015 Jul 30. PMID 26224039
- [Background] Goetze TO, Reichart A, Bankstahl US, Pauligk C, Loose M, Kraus TW, Elshafei M, Bechstein WO, Trojan J, Behrend M, Homann N, Venerito M, Bohle W, Varvenne M, Bolling C, Behringer DM, Kratz-Albers K, Siegler GM, Hozaeel W, Al-Batran SE. Adjuvant Gemcitabine Versus Neoadjuvant/Adjuvant FOLFIRINOX in Resectable Pancreatic Cancer: The Randomized Multicenter Phase II NEPAFOX Trial. Ann Surg Oncol. 2024 Jun;31(6):4073-4083. doi: 10.1245/s10434-024-15011-7. Epub 2024 Mar 8. PMID 38459418
- [Background] Gillen S, Schuster T, Meyer Zum Buschenfelde C, Friess H, Kleeff J. Preoperative/neoadjuvant therapy in pancreatic cancer: a systematic review and meta-analysis of response and resection percentages. PLoS Med. 2010 Apr 20;7(4):e1000267. doi: 10.1371/journal.pmed.1000267. PMID 20422030
- [Background] Artinyan A, Anaya DA, McKenzie S, Ellenhorn JD, Kim J. Neoadjuvant therapy is associated with improved survival in resectable pancreatic adenocarcinoma. Cancer. 2011 May 15;117(10):2044-9. doi: 10.1002/cncr.25763. Epub 2010 Nov 18. PMID 21523715
- [Background] Mokdad AA, Minter RM, Zhu H, Augustine MM, Porembka MR, Wang SC, Yopp AC, Mansour JC, Choti MA, Polanco PM. Neoadjuvant Therapy Followed by Resection Versus Upfront Resection for Resectable Pancreatic Cancer: A Propensity Score Matched Analysis. J Clin Oncol. 2017 Feb 10;35(5):515-522. doi: 10.1200/JCO.2016.68.5081. Epub 2016 Sep 30. PMID 27621388
- [Background] Lee YS, Lee JC, Yang SY, Kim J, Hwang JH. Neoadjuvant therapy versus upfront surgery in resectable pancreatic cancer according to intention-to-treat and per-protocol analysis: A systematic review and meta-analysis. Sci Rep. 2019 Oct 30;9(1):15662. doi: 10.1038/s41598-019-52167-9. PMID 31666626
- [Background] Bradley A, Van Der Meer R. Upfront Surgery versus Neoadjuvant Therapy for Resectable Pancreatic Cancer: Systematic Review and Bayesian Network Meta-analysis. Sci Rep. 2019 Mar 13;9(1):4354. doi: 10.1038/s41598-019-40951-6. PMID 30867522
- [Background] Ye M, Zhang Q, Chen Y, Fu Q, Li X, Bai X, Liang T. Neoadjuvant chemotherapy for primary resectable pancreatic cancer: a systematic review and meta-analysis. HPB (Oxford). 2020 Jun;22(6):821-832. doi: 10.1016/j.hpb.2020.01.001. Epub 2020 Jan 27. PMID 32001139
- [Background] Adam MA, Nassour I, Hoehn R, Hlavin CA, Bahary N, Bartlett DL, Lee KKW, Zureikat AH, Paniccia A. Neoadjuvant Chemotherapy for Pancreatic Adenocarcinoma Lessens the Deleterious Effect of Omission of Adjuvant Chemotherapy. Ann Surg Oncol. 2021 Jul;28(7):3800-3807. doi: 10.1245/s10434-020-09446-x. Epub 2021 Jan 1. PMID 33386547
- [Background] Birrer DL, Golcher H, Casadei R, Haile SR, Fritsch R, Hussung S, Brunner TB, Fietkau R, Meyer T, Grutzmann R, Merkel S, Ricci C, Ingaldi C, Di Marco M, Guido A, Serra C, Minni F, Pestalozzi B, Petrowsky H, DeOliveira M, Bechstein WO, Bruns CJ, Oberkofler CE, Puhan M, Lesurtel M, Heinrich S, Clavien PA. Neoadjuvant Therapy for Resectable Pancreatic Cancer: A New Standard of Care. Pooled Data From 3 Randomized Controlled Trials. Ann Surg. 2021 Nov 1;274(5):713-720. doi: 10.1097/SLA.0000000000005126. PMID 34334656
- [Background] Ghanem I, Lora D, Herradon N, de Velasco G, Carretero-Gonzalez A, Jimenez-Varas MA, Vazquez de Parga P, Feliu J. Neoadjuvant chemotherapy with or without radiotherapy versus upfront surgery for resectable pancreatic adenocarcinoma: a meta-analysis of randomized clinical trials. ESMO Open. 2022 Jun;7(3):100485. doi: 10.1016/j.esmoop.2022.100485. Epub 2022 May 14. PMID 35580504
- [Background] van Dam JL, Janssen QP, Besselink MG, Homs MYV, van Santvoort HC, van Tienhoven G, de Wilde RF, Wilmink JW, van Eijck CHJ, Groot Koerkamp B; Dutch Pancreatic Cancer Group. Neoadjuvant therapy or upfront surgery for resectable and borderline resectable pancreatic cancer: A meta-analysis of randomised controlled trials. Eur J Cancer. 2022 Jan;160:140-149. doi: 10.1016/j.ejca.2021.10.023. Epub 2021 Nov 24. PMID 34838371
- [Background] Versteijne E, Suker M, Groothuis K, Akkermans-Vogelaar JM, Besselink MG, Bonsing BA, Buijsen J, Busch OR, Creemers GM, van Dam RM, Eskens FALM, Festen S, de Groot JWB, Groot Koerkamp B, de Hingh IH, Homs MYV, van Hooft JE, Kerver ED, Luelmo SAC, Neelis KJ, Nuyttens J, Paardekooper GMRM, Patijn GA, van der Sangen MJC, de Vos-Geelen J, Wilmink JW, Zwinderman AH, Punt CJ, van Eijck CH, van Tienhoven G; Dutch Pancreatic Cancer Group. Preoperative Chemoradiotherapy Versus Immediate Surgery for Resectable and Borderline Resectable Pancreatic Cancer: Results of the Dutch Randomized Phase III PREOPANC Trial. J Clin Oncol. 2020 Jun 1;38(16):1763-1773. doi: 10.1200/JCO.19.02274. Epub 2020 Feb 27. PMID 32105518
- [Background] Pingpank JF, Hoffman JP, Ross EA, Cooper HS, Meropol NJ, Freedman G, Pinover WH, LeVoyer TE, Sasson AR, Eisenberg BL. Effect of preoperative chemoradiotherapy on surgical margin status of resected adenocarcinoma of the head of the pancreas. J Gastrointest Surg. 2001 Mar-Apr;5(2):121-30. doi: 10.1016/s1091-255x(01)80023-8. PMID 11331473
- [Background] van Geenen RC, van Gulik TM, Offerhaus GJ, de Wit LT, Busch OR, Obertop H, Gouma DJ. Survival after pancreaticoduodenectomy for periampullary adenocarcinoma: an update. Eur J Surg Oncol. 2001 Sep;27(6):549-57. doi: 10.1053/ejso.2001.1162. PMID 11520088
- [Background] Conroy T, Hammel P, Hebbar M, Ben Abdelghani M, Wei AC, Raoul JL, Chone L, Francois E, Artru P, Biagi JJ, Lecomte T, Assenat E, Faroux R, Ychou M, Volet J, Sauvanet A, Breysacher G, Di Fiore F, Cripps C, Kavan P, Texereau P, Bouhier-Leporrier K, Khemissa-Akouz F, Legoux JL, Juzyna B, Gourgou S, O'Callaghan CJ, Jouffroy-Zeller C, Rat P, Malka D, Castan F, Bachet JB; Canadian Cancer Trials Group and the Unicancer-GI-PRODIGE Group. FOLFIRINOX or Gemcitabine as Adjuvant Therapy for Pancreatic Cancer. N Engl J Med. 2018 Dec 20;379(25):2395-2406. doi: 10.1056/NEJMoa1809775. PMID 30575490
- [Background] Snyder RA, Parikh AA. Actual Survival in Patients with Resected Pancreatic Cancer: How Do Real-World Data Compare with Clinical Trial Evidence? Ann Surg Oncol. 2021 Dec;28(13):8014-8016. doi: 10.1245/s10434-021-10532-x. Epub 2021 Sep 12. No abstract available. PMID 34514521
- [Background] van Dam JL, Verkolf EMM, Dekker EN, Bonsing BA, Bratlie SO, Brosens LAA, Busch OR, van Driel LMJW, van Eijck CHJ, Feshtali S, Ghorbani P, de Groot DJA, de Groot JWB, Haberkorn BCM, de Hingh IH, van der Holt B, Karsten TM, van der Kolk MB, Labori KJ, Liem MSL, Loosveld OJL, Molenaar IQ, Polee MB, van Santvoort HC, de Vos-Geelen J, Wumkes ML, van Tienhoven G, Homs MYV, Besselink MG, Wilmink JW, Groot Koerkamp B; Dutch Pancreatic Cancer Group. Perioperative or adjuvant mFOLFIRINOX for resectable pancreatic cancer (PREOPANC-3): study protocol for a multicenter randomized controlled trial. BMC Cancer. 2023 Aug 7;23(1):728. doi: 10.1186/s12885-023-11141-5. PMID 37550634
- [Background] Labori KJ, Bratlie SO, Andersson B, Angelsen JH, Biorserud C, Bjornsson B, Bringeland EA, Elander N, Garresori H, Gronbech JE, Haux J, Hemmingsson O, Liljefors MG, Myklebust TA, Nymo LS, Peltola K, Pfeiffer P, Sallinen V, Sandstrom P, Sparrelid E, Stenvold H, Soreide K, Tingstedt B, Verbeke C, Ohlund D, Klint L, Dueland S, Lassen K; Nordic Pancreatic Cancer Trial-1 study group. Neoadjuvant FOLFIRINOX versus upfront surgery for resectable pancreatic head cancer (NORPACT-1): a multicentre, randomised, phase 2 trial. Lancet Gastroenterol Hepatol. 2024 Mar;9(3):205-217. doi: 10.1016/S2468-1253(23)00405-3. Epub 2024 Jan 15. PMID 38237621